CLINICAL TRIAL: NCT07185256
Title: A Phase 1b/2a, Open-Label, Dose-Exploration Basket Study to Investigate the Safety and Tolerability of Subretinally Injected OPGx-BEST1 Administered in Patients With Either Autosomal-Dominant BEST1 Disease (Best Vitelliform Macular Dystrophy [BVMD]) or Autosomal-Recessive Bestrophinopathy (ARB)
Brief Title: Safety and Tolerability of Subretinally Injected OPGx-BEST1 in Patients With Best Vitelliform Macular Dystrophy (BVMD) or Autosomal-Recessive Bestrophinopathy (ARB)
Acronym: BIRD-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opus Genetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPGx-BEST1 DUO-1001
Record Dates: First submitted 2025-07-17; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: ARB; BVMD; Autosomal-Dominant Bestrophinopathy; Best Vitelliform Macular Dystrophy
Keywords: Bestrophinopathy; BVMD; ARB; OPGx-BEST1; Best vitelliform macular dystrophy; Autosomal-Dominant Bestrophinopathy
MeSH Terms: conditions — Vitelliform Macular Dystrophy; Bestrophinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OPGx-BEST1 (Experimental): OPGx-BEST1, 1.5E9 vg/eye injected one time subretinally
  Interventions: Genetic: OPGx-BEST1

INTERVENTIONS:
Genetic: OPGx-BEST1 — Experimental Genetic Therapy

SUMMARY:
The goal of this clinical trial is to learn if drug OPGx-BEST1 works to treat BVMD and ARB Bestrophinopathy. It will also learn about the safety of drug OPGx-BEST1. The main questions it aims to answer are:

Evaluate the safety and tolerability of drug OPGx-BEST1 in one eye (the treatment eye), for 5 years post-injection, in participants with BVMD or ARB.

A second question it aims to answer is identification of the most appropriate dose strength of OPGx-BEST1 for clinical development.

Evaluate the efficacy of single injection of OPGx-BEST1 in one eye for 5 years post-injection.

What medical problems do participants have when taking drug OPGx-BEST1?

DETAILED DESCRIPTION:
This is a Phase 1b/2a, open-label, dose-exploring, safety and tolerability basket study of a single subretinal injection of OPGx-BEST1 in one eye of adult participants with ARB or BVMD due to BEST1 mutations.

OPGx-BEST1 has been bioengineered to include a transgene expression cassette with a codon-optimized, full-length hBEST1 gene under the control of an RPE-specific promoter. The vector genome contains inverted terminal repeats flanking an expression cassette containing the VMD2 promoter, full-length BEST1 ORF followed by SV 40 and bGH polyadenylation signal sequences, and lastly includes a kanamycin resistance gene. The Kozak sequence (upstream of the start codon) enhances the translation from the correct initiation codon. Selection of the VMD2 promoter was done to restrict the expression to the target cell type and drive expression levels comparable to those in photoreceptors. This intervention is a one-time injection.

Two vector doses are proposed for evaluation: 1.5E9 vg/eye (Cohort 1) and 4.5E9 vg/eye (Cohort 2). A minimum of 5 evaluable participants will be treated at each dose level, starting with a sentinel participant in Cohort 1. An Independent Data Monitoring Committee (IDMC) will evaluate safety 30 days after treatment of the sentinel participant before the remaining 4 participants in Cohort 1 are eligible for treatment. After the last participant has completed the Month 3 visit, the IDMC will review all Cohort 1 data and determine whether to initiate enrollment in Cohort 2 or adjust the dose escalation scheme.

Each participant will have a Screening visit and two-part Baseline visit. On Day 1 (Visit 4), participants will undergo vitrectomy with subretinal injection of OPGx-BEST1 at the preassigned dose. Participants will return for follow-up on Day 2, Day 7, Day 14, Day 30, and Day 45 following IMP administration (Visits 5-9). Participants will also return 3 and 6 months following IMP administration (Visits 10-11) and 1, 1.5, 2, 3, 4, and 5 years following IMP administration (Visits 12-17).

Post-IMP administration, safety and efficacy outcomes will be evaluated for 5 years.

In addition to the primary objectives of establishing IMP safety and tolerability and identifying the most appropriate dose strength, the study will evaluate the preliminary efficacy of OPGx-BEST1 and characterize the immunogenic effects of administration. A central reading center will provide standardized evaluation of select imaging data. Analysis of results will include treatment-eye comparisons of visual function post-administration of OPGx-BEST1 to baseline visual function.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all the following criteria will be eligible to participate in the study:

1. Provide informed consent to study assessments.
2. Able and willing to comply with all study assessments for the duration of the study.
3. ≥18 years old.
4. ETDRS BCVA measured with standard testing distances:

   1. For the sentinel participant in each cohort, ≤20 letters (Snellen equivalent of 20/200 [1.30 logMAR] or worse)
   2. For subsequent participants in the same cohort, 65 to 20 letters inclusive (Snellen equivalent of 20/50 [0.40 logMAR] to 20/200 [1.30 logMAR]).
5. Genetic confirmation on chromosome 11q12-q13.1 of BVMD or ARB with a BEST1 genetic test or IRD panel test including a BEST1 variant test, by a Clinical Laboratory Improvement Amendments (CLIA) or European certified laboratory. If available test result is more than 15 years old, confirmation testing will be performed at Visit 1, with results needed by Visit 3.
6. Confirmation of one disease-causing (pathogenic or likely pathogenic, autosomal-dominant) variant in the BEST1 gene for BVMD, as listed in the IB, or two variants for ARB per American College of Medical Genetics and Genomics/Association for Molecular Pathology (ACMG/AMP) variant interpretation.
7. BVMD: Clinical phenotype and diagnosis consistent with advanced BVMD with active subretinal fluid or vitelliform material.
8. ARB: Clinical phenotype and diagnosis consistent with ARB.

Exclusion Criteria:

Individuals who meet any of the following criteria will not be eligible to participate in the study.

1. Women of childbearing potential (WOCBP) who are pregnant, lactating, and/or unwilling to use effective contraception from Screening through 1 year after IMP administration. See Section 13.3 (Appendix 3) for contraception guidelines.
2. Men who are unwilling to use adequate contraception from Screening through 180 days after IMP administration. See Section 13.3 (Appendix 3) for contraception guidelines.
3. Have a pre-existing eye condition or complicating systemic disease that could preclude the planned surgery (e.g., individuals who are immunocompromised, on continuous systemic immunosuppressive treatment or anticipate a need to initiate it for non-study reasons, or unable to take the concomitant immuno-suppressive regimen necessary for IMP administration).
4. Have a history of disease that may preclude the individual from study participation (e.g., other bestrophinopathy, such as AOFVD or ADVIRC) or that may interfere with or preclude outcome measure testing as described in the protocol.
5. Have previously received gene therapy of any kind.
6. Presence of active choroidal neovascularization (CNV) that, in the opinion of the Investigator, affects vision or may require treatment.
7. Presence of subretinal fibrosis that may significantly limit improvement in visual acuity.
8. Have an epiretinal membrane that may require surgical intervention.
9. Have undergone tube surgery for glaucoma at any time or have glaucoma that has been unstable within the past 4 years. Note: Prior incisional surgery (e.g., trabeculectomy and iridotomy) is not exclusionary.
10. Had intraocular surgery within 90 days prior to planned IMP administration or have active inflammation at Screening resulting from prior ocular surgery.
11. Have used any investigational drug or device within 90 days prior to planned IMP administration or plan to participate in another drug or device study during the same period as the current study.
12. Have received a vaccination within 6 weeks prior to planned IMP administration or plan to be vaccinated within 6 months after IMP administration.
13. Have received anticoagulant therapy within 2 weeks prior to planned IMP administration.
14. Have active macular neovascularization as determined by OCT-A.
15. Are incapable of performing visual function testing for reasons other than poor vision.
16. Have any contraindication to the concomitant steroid regiment proscribed in the protocol.
17. Have any other condition (ocular, medical, or psychological) that would not allow the individual to complete follow-up examinations during the study and/or, in the opinion of the Investigator, makes it hazardous or unsuitable for the individual to participate in the study.
18. Have a known history of hypersensitivity to constituents or excipients in the pharmaceutical formulation of the IMP.
19. Have a known infection of human immunodeficiency virus (HIV), hepatitis B or C virus, or herpes simplex virus.
20. Are an employee of the Sponsor or a relative of the Investigator or investigative site staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicity (DLT) events at the dose tested | 5 years
  Number of dose-limiting toxicity (DLT) events, defined as any ≥Grade 3 toxicity that occurs within 90 days after IMP administration based on the National Cancer Institute common toxicity criteria
Number and severity of procedure-related adverse events | 5 years
  Number and severity of adverse events related to the administration of OPGx-BEST1 involving pars plana vitrectomy and subretinal injection under general anesthesia
Number and severity of adverse events related to OPGx-BEST1 | 5 years
  Number and severity of adverse events considered related to the study drug, OPGx-BEST1

SECONDARY OUTCOMES:
Changes from baseline in retinal morphology assessed by spectral-domain optical coherence tomography | 5 years
  Changes from baseline in retinal morphology assessed by spectral-domain optical coherence tomography
Changes from baseline in retinal morphology assessed by 55 degree fundus autofluorescence (FAF) | 5 years
  Changes from baseline in retinal morphology assessed by 55 degree fundus autofluorescence (FAF)
Changes from baseline in retinal morphology assessed by ultra-wide angle autofluorescence (FAF) | 5 years
  Changes from baseline in retinal morphology assessed by ultra-wide angle autofluorescence (FAF)
Changes from baseline in neovascularization assessed by optical coherence tomography | 5 years
  Changes from baseline in neovascularization assessed by optical coherence tomography angiography
Changes from baseline in retinal sensitivity | 5 years
  Changes from baseline in retinal sensitivity assessed by microperimetry
Changes from baseline in best corrected visual acuity | 5 years
  Changes from baseline in best corrected visual acuity letter score as measured by Early Treatment Diabetic Retinopathy Stuidy (ETDRS) charts
Changes from baseline in low luminance visual acuity | 5 years
  Changes from baseline in low luminance visual acuity assessed by ETDRS charts
Changes from baseline in participant-reported outcomes | 5 years
  Changes from baseline in participant-reported outcomes assessed by the Michigan Retinal Degeneration Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Opus website with description of programs — https://opusgtx.com/pipeline-programs/